# 广东医科大学附属医院临床研究

# 申请书

申报类型:[]大型队列研究 []重点项目 [√]一般项目

改良 Blumgart 对比传统 Blumgart 的胰肠吻合技术项目名称: 在腹腔镜胰十二指肠切除术治疗壶腹周围癌对术后 胰瘘的影响: 一项开放、随机、平行对照临床研究

申请者: 刘国华

所在科室: 肝胆胰外科

联系电话: 13659791525

电子信箱: lgheagle@126.com

版本号: 4.0

版本日期: 2023.6.30

广东医科大学附属医院临床研究中心

二〇二一年制

## 一、科室意见

## 申请者承诺

我保证本申请书填报内容的真实性。如果获得资助,我与本项目组成员将严格遵守《广东医科大学附属医院临床研究管理办法(试行)》的有关规定,切实保证研究工作时间,按计划认真开展研究工作,按时报送有关材料。

申请者(签章)

年 月 日

## 科室意见

科主任(签章):

年 月 日

## 二、基本信息

| 申 | 姓 名 | 刘国华 | 性别 | 男 | 出生年月 | 1977年8月 | 民族 | 汉族 |
|---|---|---|---|---|---|---|---|---|
| 请 | 职 称 | 主任医师 | 主任医师 | | | 肝胆胰外科 | | |
| 人 | 学 位 | 硕士 | 硕士 | | 授予年份 | 2012 年 | | |
| 信 | 电 话 | 1365979152 | 25 | | 电子邮箱 | lgheagle@126.com | | |
| 息 | 主要研究<br>领域 | 肝胆胰的基础 | 肝胆胰的基础与临床研究 | | | | | |
| 项目 | 项目名称 | 改良 Blumgart 对比传统 Blumgart 的胰肠吻合技术在腹腔镜胰十二指肠切除术治疗壶腹周围癌对术后胰瘘的影响:一项开放、随机、平行对照临床研究 | | | | | | |
| 基本信息 | 研究类型 | []队列研 | [√]临床试验(随机对照试验) [ ]病例对照研究 [ ]横断面研究 [ ]诊断性研究 [ ]其它 (请在最符合的一个研究类型前打"√") | | | | | |
| <b>研究年限</b> 2023 年 8 月至 2028 年 8 月 <b>申请经费</b> | | | | 2: | 5 万元 | | | |

摘要(500字以内

壶腹周围癌在国内外的发病率和病死率均显现出上升趋势,严重影响人民的健康水平。实施胰十二指肠切除术(PD)是壶腹周围癌唯一有效的治疗措施,但是由于PD 手术的技术复杂、困难,而腹腔镜胰十二指肠切除术(LPD)难度更大,且术后死亡率可达 5%,其重要原因是出现最严重的并发症一胰瘘。胰瘘的发生与众多因素相关,最关键也是术者可以掌控的因素是胰肠吻合的方式和技术,所以胰肠吻合技术的改进创新一直是外科临床研究的热点。Blumgart 胰肠吻合技术最初是由美国 L. H. Blumgart 教授所创的,因其较低的胰瘘发生率而得以在 OPD 中被广泛应用,但传统的 Blumgart 吻合步骤繁杂,并不适宜在 LPD 中应用。而本团队根据自身的经验对传统 Blumgart 吻合进行简化改良后应用于 OPD 并通过回顾性研究发现其除了具备操作简便的特点外、还具有较低胰瘘发生率的优势,然而,在 LPD 中的应用价值仍需进一步探讨。因此,本研究拟采用前瞻性随机对照试验,将行传统 Blumgart 胰肠吻合的 LPD 患者作为对照组,将本团队设计改良 Blumgart 胰肠吻合的 LPD 患者作为对照组,将本团队设计改良 Blumgart 胰肠吻合的 LPD 患者作为对照组,将本团队设计改良 Blumgart 胰肠吻合的 LPD 患者作为对照组,通过对比两组患者的临床相关指标及术后并发症发生率,探讨该技术在 LPD 中的应用价值即能否真正做到简化手术步骤的同时保证较低的胰漏发生率。

关键词

腹腔镜胰十二指肠切除术、胰腺瘘、Blumgart 吻合术、壶腹周围癌

## 三、项目组人员(含主要研究者)

| 姓名 | 单位 | 学位 | 职称 | 项目任务 | 伦理培训 | GCP 培训 | 签名 |
|-----|-------|----|------|----------------|------|--------|----|
| | | | | 分工 | | | |
| 刘国华 | 广东医科大 | 硕士 | 主任医师 | 课题负责 | 有 | 有 | |
| | 学附属医院 | | | 人 | | | |
| 李明意 | 广东医科大 | 博士 | 教授 | 项目指导 | 有 | 有 | |
| | 学附属医院 | | | | | | |
| 谭小宇 | 广东医科大 | 学士 | 主任医师 | 项目实施、 | 有 | 有 | |
| | 学附属医院 | | | 病例的观<br> 察,随访 | | | |
| 吴家园 | 广东医科大 | 博士 | 副主任医 | 数据整理、 | 有 | 有 | |
| | 学附属医院 | | 师 | 统计分析 | | | |
| 钟国辉 | 广东医科大 | 硕士 | 住院医师 | 项目实施、 | 无 | 有 | |
| | 学附属医院 | | | 病例的观<br> 察,随访 | | | |
| 翟景威 | 广东医科大 | 硕士 | 住院医师 | 项目实施、 | 无 | 无 | |
| | 学附属医院 | | | 病例的观<br> 察,随访 | | | |
| 邓春梅 | 广东医科大 | 本科 | 副主任护 | 病例随访、 | 无 | 无 | |
| | 学附属医院 | | 师 | 记录 | | | |
| 许俊儿 | 广东医科大 | 本科 | 主管护师 | 病例随访、 | 无 | 无 | |
| | 学附属医院 | | | 记录 | | | |
| 李嘉兴 | 广东医科大 | 硕士 | 住院医师 | 项目数据 | 无 | 无 | |
| | 学附属医院 | | | 的收集、分<br> 析 | | | |
| 钟瑜 | 广东医科大 | 硕士 | 住院医师 | 项目实施、 | 无 | 无 | |
| | 学附属医院 | | | 病例的观<br>察,随访 | | | |
| 徐振越 | 广东医科大 | 硕士 | 规培医师 | 病例的观 | 无 | 无 | |
| | 学附属医院 | 在读 | | 察,随访 | | | |

项目秘书: 翟景威 联系方式: 18814103880 邮箱: 466269963@qq.com

#### 四、申请者工作积累

- 1.申请人临床工作中有丰富的经验积累,本项目开展所需的相关技术储备充分:
- (1)本人自2002年起一直从事于肝胆胰外科专业至今已有20余年,临床相关专业经验丰富。现任广东省医学会外科学分会肝胆胰分会肝脏学组委员、广东省抗癌协会胰腺癌专业青年委员会常务委员、广东省健康管理学会肝胆胰专业委员会常务委员、湛江市医学会微创外科分会常务委员等多个专业学会任职。
- (2)本项目开展所需的相关技术储备充分: 2016 年聘任副主任医师后便确定以胆胰微创治疗等临床研究作为专业研究方向。2017 年到浙江省人民医院胆胰微创中心进修学习腹腔镜胰十二指肠切除术(LPD)相关技术,回来后协助我科学科带头人李明意教授、谭小宇教授筹建了我院胆胰亚专科中心,并取得了不少荣誉和成绩: 如 2018 年开展新技术 LPD 并帮助本团队获得医院的新技术奖,成功开展湛江市首例 LPD;并将本团队独创的改良 Blumgar 胰肠吻合技术应用于 LPD中。2019 年、2020 年连续两年受邀出席广东省医学会肝胆胰学术会议介绍了相关技术工作。在 2019 年参加广东省肝胆胰手术视频大赛获得季军,2021 年参加全国华南肝胆胰手术视频大赛获得二等奖。目前我胆胰胆胰亚专科中心已能常规开展高难度胰腺相关微创手术:如腹腔镜胰体尾(保留脾脏)切除术(Kimura 法或 Warshaw 法);腹腔镜胰体尾癌根治性切除术(RAMPS);腹腔镜胰十二指肠切除术(LPD)等。
- 2. 申请人有丰富的临床研究和基础研究经验,并已有开展本项目前期技术相关的研究基础:
- (1)参与或主持国家级、省、市级课题项目
  - ①2009 年 国家自然基金项目 《维生素 K2 通过 SXR 调控 Matrilin-2 促进卵圆细胞 增殖介导肝再生的研究》(参与人)。
  - ②2011年 省自然基金项目《SXR在 matrilin-2 促进卵圆细胞增殖介导肝再生中调控作用的研究》(第三完成人)。
  - ③2018 年 湛江市科技项目《湛江市地区胆石症患者术中胆汁菌群分布、药敏分析临床研究》(项目负责人)。
- (2)发表多篇胆胰专业领域相关临床研究论文,其中前两篇是与本项目密切相关的胰腺手术技术的临床研究论文。
  - (1) SCI: Liu G, Tan X, Li J, Zhong G, Zhai JandLi M(2022). Casereport: Treatment of intraductal Papillary mucinous neoplasms located in middle-segment pancreas with end-to-end anastomosis reconstruction after laparoscopic central pancreatectomy surgery through a pigtail-tube-stent placement of the pancreatic duct. Front. Surg. 9:937682.doi:10.3389/fsurg.2022.937682.
  - ②中文核心: 刘国华, 谭小宇, 戴东, 等. 改良 Blumgart 胰肠吻合在胰十二指肠切除术中的应用[J]. 中国普通外科杂志, 2020, 29(3):276-283.
- ③中文核心: 刘国华, 谭小宇, 戴东, 等. 循 PCD 引流管路径微小切口联合经皮肾镜治疗重症急性胰腺炎感染性坏死. 中国普通外科杂志. 2018. 3. 335-342.
- ④中文: 刘国华, 刘架形, 谭小宇, 等. 急性胆管炎患者胆汁培养结果和药敏分析. 岭南现代临床外科. 2020. 20(1):29-33.
  - (5)中文: 刘国华, 谭小宇, 戴东, 等. 利胆排石方在胆石术后胆道镜探查取石的临床应

| 用分析. 齐齐哈尔医学院学报. 2 | 2013. 13. 1033–1034. |
|-------------------|----------------------|

## 五、创新性和可行性分析

#### 1. 本项目特色及创新性

本研究在以往回顾性研究基础上,采用前瞻性随机对照实验,设置对照组实验,将行传统 Blumgart 胰肠吻合的 LPD 患者作为对照组,将本团队设计改良 Blumgart 胰肠吻合的 LPD 患者作为试验组,通过对比两组患者的临床相关指标及术后并发症发生率,探讨本团队设计改良 Blumgart 胰肠吻合在 LPD 术中的应用效果以及安全性。该胰肠吻合术式是笔者团队在多年的普外科手术经验以及深入了解各种胰肠吻合方式的基础上对 Blumgart 胰肠吻合的复杂步骤进行简化、改良所得出的,目前在国内外文献报道中均未发现同类型吻合方式的相关研究。

2. 可行性分析(科室条件、人员配备、病例来源、技术条件等)

广东医科大学附属医院是粤西地区规模最大综合型"三级甲等医院",是区域内唯一一家集医疗、教学、科研、预防保健为一体的大型医学中心。医院先后获得广东省首批三级甲等医院、全国文明单位、全国"百佳"医院、全国巾帼文明示范岗等荣誉称号 120 多项。广东医科大学附属医院肝胆外科在粤西地区具有极高的影响力。

本团队前期在改良 Blumgart 胰肠吻合在 LPD 术中的应用效果以及安全性的研究中已积累一定的临床经验,在 2020 年回顾性分析研究中,本团队将 2014 年 8 月-2017年1月 55 例 PD 术中采用传统空肠套入式胰肠吻合的患者(传统组)与 2017年2月-2019年 8 月 53 例 PD 术中采用改良 Blumgart 胰肠吻合的患者进行对照研究,通过比较两组

患者的相关临床指标以及术后并发症发生率,发现 PD 术中采用改良 Blumgart 胰肠吻合可有效降低术后胰瘘、腹腔出血、腹腔感染并发症的发生率,并且把该研究结果以论文的形式发表在中国普通外科杂志。

根据相关报道指出,壶腹周围癌在国内外的发病率均显现出上升趋势,在粤西地区范围内也有着相同的趋势,因此,需要行胰十二指肠切除术的患者也越来越多。本研究团队目前拥有高级职称技术人员3人(李明意教授、谭小宇教授、刘国华教授),已成功实施多台腹腔镜胰十二指肠切除术,在保证手术成功率的同时亦能从容应对各种术后并发症;住院医师2人(均为硕士及以上学历),具有丰富的患者随访及统计分析经验,能保证临床数据记录以及统计分析的准确性,人才梯度合理,分工明确,能保证本课题的顺利完成。

## 六、进度计划和预期目标

1. 进度计划(包括各年度任务目标、考核指标及研究开发内容完成的计划进度。按年度进行填写,每年度的研究计划和目标应明确、可考核,并能与课题整体研究任务、完成时间、考核指标相对应。)

2023.08-2024.07 ①成功入组 34 例 LPD 患者(进行随机化分组,术中采用传统 Blumgart 胰肠吻合 or 改良 Blumgart 胰肠吻合),收集患者 相关临床指标及术后并发症发生情况,并对数据进行系统记录

2024.08-2025.07 ②成功入组 34 例 LPD 患者 (进行随机化分组, 采用传统 Blumgart 胰肠吻合), 其余同上

## 广东医学院附属医院临床研究课题申请书

2028.04-2028.08 (7)攥写论文。

- 2. 预期目标与考核指标(重点说明本研究完成的最终成果和载体形式,如论文、成果、专利等;考核指标内容需完整、明确,能够考查课题完成的程度和实际效果。)
- (1) 探究改良 Blumgart 胰肠吻合在腹腔镜胰十二指肠切除术中的应用效果及安全性
- (2) 发表与临床研究相关的 SCI 文章 1 篇。

### 七、经费预算

| 序号 | 预算科目名称 | 经费预算(万) | 备 注<br>(计算依据与说明) |
|----|-------------|---------|-----------------------------------------------|
| 1 | 临床研究业务费 | 6 | 计划书、CRF表的制定费,研究助理及研究者培训费,研究生劳务费、外出学习、文献检索等费用。 |
| 2 | 咨询费、调研费和劳务费 | 10 | 专家咨询费、论文发表,润色、<br>入组病例调查随访费等 |
| 3 | 资料费 | 2 | 复印打印费,资料统计分析费等。 |
| 4 | 协作费 | 5 | 课题实施过程中需要协作或调 研所支付的费用。 |
| 5 | 交通费 | 2 | 外出学习交通费 |
| | 合计 | 25 | |

改良 Blumgart 对比传统 Blumgart 的胰肠吻合技术在腹腔镜胰十二指肠切除术治疗壶腹周围癌对术后胰瘘的影响:

一项开放、随机、平行对照临床研究

# 研究方案

研究负责人: 刘国华主任医师

申办方:广东医科大学附属医院

版本号: 4.0

版本日期: 2023-6-30

## 目录

| 方 | 案摘要 <del></del> |
|----|--------------------------------------------------------------------|
| 1. | 研究背景(立项依据)———————— |
| | 参考文献 |
| 2. | 研究目的 ———————————————————————————————————— |
| 3. | 研究对象 ———————————————————————————————————— |
| | 3.1 入选标准———————————————————————————————————— |
| | 3.2 排除标准———————————————————————————————————— |
| | 3.3 退出标准 |
| 4. | 方案设计 |
| 5. | 样本量计算及分组 |
| | 5.1 样本量估算 |
| | 5.2 患者编号和随机化分组 ———————————————————————————————————— |
| 6. | 研究步骤(治疗方案)———————————————————————————————————— |
| | 6.1 术前筛查 ———————————————————————————————————— |
| | 6.2 手术方案 ———————————————————————————————————— |
| | 6.2.1 试验组及对照组共同的 LPD 手术流程 ———————————————————————————————————— |
| | 6.2.2 试验组的改良 Blumgart 胰肠吻合的方案 ———————————————————————————————————— |
| | 6.2.3 对照组的传统 Blumgart 胰肠吻合的方案 ———————————————————————————————————— |
| | 6.3 手术人员要求 — 1 |
| | 6.4 术后治疗方案 |
| | 6.5 手术后出院标准 ———————————————————————————————————— |
| 7. | 随访方案 |
| 8. | 研究结果评价指标及方法 |
| | 8.1 主要指标 ———————————————————————————————————— |
| | 8.2 次要指标 ———————————————————————————————————— |
| 9. | 安全性评价 ———————————————————————————————————— |
| | 9.1 获益 ——————————————————————————————————— |

| 9.2 风险 ——————————————————————————————————— | <b>-</b> 15 |
|--------------------------------------------------------|-------------|
| 9.3 风险防范措施———————————————————————————————————— | <b>-</b> 15 |
| 9.3.1 指导原则 ———————————————————————————————————— | <b>-</b> 15 |
| 9.3.2 组织管理 ———————————————————————————————————— | <b>-</b> 16 |
| 9.3.3 防范措施 ———————————————————————————————————— | <b>–</b> 16 |
| 9.3.4 不良事件 | <b>–</b> 17 |
| 9.3.4.1 严重不良事件的定义 ———————————————————————————————————— | |
| 9.3.4.2 因果关系 ———————————————————————————————————— | <b>-</b> 18 |
| 9.3.4.3 预期不良事件 ———————————————————————————————————— | <b>-</b> 19 |
| 9.3.4.4 不良事件处理措施 ———————————————————————————————————— | <b>-</b> 19 |
| 9.3.5 突发事件处理措施 ———————————————————————————————————— | <b>-</b> 20 |
| 9.3.6 处罚 ——————————————————————————————————— | <b>-</b> 21 |
| 10.招募过程 | <b>-</b> 21 |
| 10.1 招募程序 ———————————————————————————————————— | • 21 |
| 10.2 启动时间 ———————————————————————————————————— | - 22 |
| 10.3 招募材料 ———————————————————————————————————— | <b>-</b> 22 |
| 10.4 预期招募人数 ———————————————————————————————————— | <b>2</b> 2 |
| 10.5 研究对象参加研究的时间 ———————————————————————————————————— | <b>-</b> 23 |
| 11.数据管理与统计分析计划 ———————————————————————————————————— | <b>-</b> 23 |
| 12. 资料保密计划 ———————————————————————————————————— | <b>-</b> 24 |
| 13.伦理要求与知情同意 | <b>-</b> 25 |
| 14.质量控制和质量保证 ———————————————————————————————————— | <b>-</b> 26 |
| 15.数据和记录的保存 ———————————————————————————————————— | <b>-</b> 26 |
| 16.研究流程 ———————————————————————————————————— | <b>-</b> 27 |
| 附录: ———————————————————————————————————— | 28-39 |

附录 1. 试验流程

附录 2. 评估时间表及流程

附录 3. ASA 分级标准

附录 4. ECOG 体力状态评分标准

附录 5. 随机化申请表

附录 6. AJCC 壶腹癌分期标准(2018年第八版)

附录 7. ISGPS 术后胰瘘 (POPF) 定义及分级标准 (2016 版)

附录 8. 术后并发症 Clevieu-Dindo 系统分级

附录 9. 国际生命质量(EORTC QLQ C30)问卷

## 方案摘要

| 研究名称 | 改良 Blumgart 对比传统 Blumgart 的胰肠吻合技术在腹腔镜胰十二指 |
|---|---|
| -917 <b>3</b> H 14. | |
| | 对照临床研究 |
| → ਜਜ <i>ਹ</i> ੁਹ <del>ਲੋ ਂ</del> . | V |
| 主要研究者 | 刘国华主任医师 |
| 研究目的 | 以腹腔镜下传统 Blumgart 胰肠吻合术作为对照,评价探讨本团队设计 |
| | 改良 Blumgart 胰肠吻合术在 LPD 中的应用价值即能否真正做到简化手 |
| | 术步骤的同时保证较低的胰漏发生率。 |
| 主要评价指标 | 术后胰瘘发生率(POPF) |
| (疗效指标) | |
| 次要评价指标 | 围手术期安全性 |
| (疗效指标) | 胰肠吻合所耗费时间(PJ-time) |
| | LPD 手术总耗费时间 |
| | 术中出血量 |
| | 术中中转率 |
| | 术后 30 天内除胰瘘外其他主要并发症发生率 |
| | (腹腔感染、腹腔出血、胃排空延迟) |
| | 术后恢复情况 |
| | 术后疼痛评分 |
| | 术后首次排气时间 |
| | 术后开始进食时间 |
| | 住院天数 |
| | 术后生活质量 |
| | 生活质量评分 (EORTC QLQ C30 问卷) |
| 次要评价指标 | 术后 90 天内死亡率 |
| (安全性指标) | |

# 1) 年龄 18-80 岁; 入选标准 2) 影像学(上腹部MRI、MRCP/CT/CTA)诊断为壶腹周围(十二指肠乳 头、壶腹部、胆总管下段、胰头部)肿瘤性病变; 3) 经MDT讨论评估肿瘤未侵犯大血管(SMA,CA,CHA/SMV,PV) 可切 除; 4) 十二指肠超声内镜下诊断为壶腹周围癌; 5) 内镜下活检病理证实为癌(非必需); 6) 术前分期为 T3N1 以内: 7) 未发现远处转移证据者: 8) 心肺及肝肾功能可耐受手术; 9) 患者及家属能够理解并愿意参与本研究,提供书面知情同意。 排除标准 1) 诊断合并其他部位恶性肿瘤; 2) ASA分级 ≥ IV级和/或ECOG体力状态评分> 2分: 3) 具有严重的肝肾功能、心肺功能、凝血功能障碍或合并严重的基础 疾病不能耐受手术者; 4) 术前有感染未控制者; 5) 怀孕或哺乳期妇女; 6) 具有严重的精神疾病病史; 7)有研究者认为的其他临床、实验室情况病人不宜参加该项试验。 退出标准 1) 术中探查证实远处转移患者,包括肝脏、盆腔、腹膜等; 2) 术中探查证实肿瘤无法根治性切除,需要改行姑息性短路手术如: 胆肠吻合的患者: 3) 术中因各种因素导致手术中转开腹或终止手术的患者。 4)入选研究后,患者因各种原因要求退出本研究队列者; 5)入选研究后因各种原因患者不能或不愿继续完成研究计划者。

## 受试者数量

样本量验证

计划入选患者例数为 150 例,实验组与对照组均为 75 例。

预计所有受试者招募入组时限为4年左右,术后随访时限为90天。本研究为平行对照设计的临床研究,试验组为采取改良Blumgart吻合的LPD患者,对照组为采取传统Blumgart吻合的LPD患者,观察试验组患者术后POPF发生率是否低于对照组患者。根据既往文献报道以及本团队既往手术经验:估计试验组的术后POPF发生率约为6%,对照组的术后POPF发生率约为16%,试验组与对照组按1:1比例分组,按照优效性试验两组总样本率计算,优效界值 $\triangle$ =5%, $\alpha$ =0.05, $\beta$ =0.2(功效=80%),利用PASS11软件计算得到试验组和对照组所需要的最小样本量 $N_1$ = $N_2$ =67 例,假定研究对象的失访率为10%,则需要样本量 $N_1$ = $N_2$ =67÷0.9 $\approx$ 75例,即总样本量为150例。

#### 治疗方案

#### 1. 手术方案:

符合入选标准的患者,接受随机化分组后,分别进行改良 Blumgart 吻合的 LPD 手术或传统 Blumgart 胰肠吻合的 LPD 手术;

### 2. 术后治疗方案:

术后予以术后抗感染、护肝、营养支持和抑制胰液分泌等治疗,抑制胰液分泌的药物治疗方案选择以生长因素或类似物方案。

### 1. 立题依据

壶腹周围癌在国内外的发病率显现出上升趋势,据相关报道<sup>[11</sup>指出,壶腹周围癌发病率在恶性肿瘤中居第 8~9 位,但病死率却高居肿瘤的第 4 位,严重影响人民的健康水平。而实施胰十二指肠切除术(pancreaticoduodenectomy,PD)是其唯一有效的治疗措施。1953年,外科医师 Whipple 首次开创胰十二指肠切除术,后来该术式被广泛应用<sup>[2]</sup>。直至目前,PD 仍是壶腹周围癌及胰头癌的标准术式,因其切除范围广,解剖关系复杂、吻合技术困难、且并发症发生率高,曾被誉为普通外科手术"王冠上的明珠"。因此,尽管微创外科迎来蓬勃的发展,其在 PD 术中的应用却相对落后。直至 1994年,Gagner 和 Pomp<sup>[3]</sup>首次报道腹腔镜胰十二指肠切除术(laparoscopic pancreaticoduodenectomy,LPD),初步验证了其在该领域的安全性以及可行性,但与传统开放式胰十二指肠切除术(Open pancreaticoduodenectomy,OPD)相比,LPD 对于术者的技术要求则更高,例如二维视觉、手术器械自由活动度以及手眼协调性、操作精准性等,所以 LPD 也被称为微创外科中的"珠穆朗玛峰"。近年来,随着网络媒体的快速发展以及 3D 腹腔镜的投入使用,外科医生可通过线上学习和会议交流来缩短学习曲线,精进操作技术,改良手术方案;同时 3D 视觉也使得解剖分离、吻合层次变得更加清晰,突破了切除吻合困难这个瓶颈,使普通外科医师们能够征服 LPD 这座"珠穆朗玛峰"。

要想征服 LPD 这座"珠穆朗玛峰",胰瘘这一术后并发症是所有普通外科医师都必须解决的难题。术后胰瘘与众多因素相关,例如年龄、BMI、肿瘤类型、胰腺质地、胰肠吻合的方式与技术<sup>[4]</sup>等等,但其中最关键也是操作者唯一可以改变的因素则是胰肠吻合技术。因此胰肠吻合方式的创新一直是研究热点。自 Whipple 开创 PD 手术方式以来,术中标本切除后的胰腺连续性重建主要有两种方式: 胰肠吻合、胰胃吻合。这两种重建方式哪种更有优势? 国外的多项随机对照研究<sup>[5-7]</sup>表明 ,胰肠吻合和胰胃吻合在术后胰瘘发生率上并无显著性差异。尽管如此,来自 ISGPS 的一项调查<sup>[8]</sup>显示 : 超过 80%的外科医生在 OPD或 LPD 中均选择了胰肠吻合。所以,目前胰肠吻合仍是胰腺连续性重建的主流方向,而围绕着胰肠吻合技术的各种改进方法层出不穷,这就不难明白虽然胰肠套入式吻合与胰管空肠黏膜吻合是胰肠吻合的两种主要方式<sup>[9]</sup> ,但吻合方法却多达 50 余种这其中的道理了。

那么,LPD 中胰肠吻合的方式及方法该如何选择呢?其实目前的国内外研究仍然没有达成共识。

首先,胰肠套入式吻合是将胰腺断端完全套入至空肠腔使胰液导入空肠腔理论上减少了胰液向吻合口外渗漏,但早期胰肠套入式吻合忽视了胰液进入空肠后激活胰酶对吻合口的影响导致吻合口瘘甚至出血等严重后果。尽管后期也有相关研究提示某些胰肠套入式吻合方法也能获得较低胰漏发生率,譬如:2007年彭淑牖等[10]报道的捆绑式胰腺套入吻合法和陈孝平等[11]近年来提出的陈氏 U 型套人缝合法。但是就本团队前期回顾性研究[11]中,对照组采用的就是较为传统的胰肠套入式吻合方法,所取得的效果并不理想,在 55 例的患者中就有 10 例发生了 B/C 级胰瘘,胰瘘的发生率高达 18.8%,同时发生腹腔出血 8 例,死亡4 例,死亡原因均为胰瘘导致的腹腔出血引起。分析其原因,本团队实施的传统胰肠套入式吻合方法虽然在胰腺断面套入空肠前已通过一支架管置入主胰管将胰液导入空肠并尽可能使它远离胰肠吻合口,但由于套入前并未对胰腺断面进行预处理其实还是忽视了胰腺断面副胰管的存在,同时,套入式吻合本身难以避免的将胰腺断面裸露在空肠腔内,这就为胰酶的激活等一系列反应创造了条件,胰瘘和吻合口出血乃至腹腔出血发生的概率便更高了。另外,由于上述胰肠套入式吻合方法在腹腔镜下对操作的要求更高,步骤复杂,难以理解,故而在 LPD 中应用并不多。

其次,胰管空肠黏膜吻合方式则是将主胰管与空肠作黏膜对黏膜的缝合,这样做除了能将胰液导入空肠腔内以外,还将胰液与胰腺断面与空肠黏膜完全隔离,从而减少了胰液对吻合口的影响,理论上应该能极大减少胰漏提高 PD 的安全性。但由于早期胰管空肠黏膜吻合仍然忽视了胰腺断面副胰管的存在,断面的胰液渗漏淤积在胰腺空肠浆膜之间的间隙从而形成死腔,故效果并不理想。2010 年美国 Blumgart 教授报道了关于 Blumgart 胰管空肠黏膜吻合技术研究并指出该吻合方法是通过贯穿胰腺全层与空肠浆肌层的间断褥式缝合,可有效降低缝线对胰腺组织的剪切力,同时能保证空肠浆膜面 对胰腺断面的有效覆盖,避免死腔形成<sup>[12]</sup>,因而可明显降低术后胰瘘等术后并发症发生率。而传统的 Blumgart 吻合操作步骤相对复杂,一开始并未被广泛应用。此后出现了各种改良 Blumgart 吻合方法并应用于 OPD 手术中,多项研究[13-16] 也指出 Blumgart 吻合或者改良 Blumgart 吻合为手术步骤中均要进行多针的空肠与胰管的黏膜对黏膜缝合,这对较小胰管的胰肠吻合来说在腹腔镜下操作更难,因此,该技术难以在 LPD 中推广。目前 PubMed,EMBASE 和 Cochrane databases 搜索有关 Blumgart 吻合

在 LPD 应用的临床研究仅有几篇[7, 17-18], 且均属于回顾性研究。

综上所述,如能设计一种更为简单易于操作且兼具较低胰漏发生率的改良 Blumgart 吻合将利于 Blumgart 胰肠吻合推广应用于 LPD, 进一步造福人民的健康。而本技术团队在前期设计了一种简易 Blumgart 吻合并将其应用于 OPD 中并取得了较好的手术效果,其改良方案是:胰管支撑管与主胰管用荷包缝合的方法充分固定后通过空肠黏膜戳孔处置入空肠腔后再作一荷包缝合关闭戳孔与支撑管间隙,理论上主胰管的胰液渗漏会更低且减少了胰管黏膜吻合这一繁琐的步骤;而贯穿胰腺全层与空肠浆肌层的间断交锁缝合能有效防止副胰管胰液渗漏,同时胰腺前壁与空肠浆肌层的间断交锁 U 型缝合能使空肠浆膜面对胰腺断面的有效覆盖更加严密,避免死腔形成。当然,由于之前的研究仅仅应用于 OPD 中,属于回顾性研究且样本量偏少,病例选择亦可能存在偏倚。因此,对于经本技术团队改良的这一简易 Blumgart 胰肠吻合技术的临床应用价值需要通过前瞻性随机对照的临床研究作进一步评价。

基于上述原因,本胆胰亚专科中心拟通过开展"腹腔镜胰十二指肠切除术应用改良 Blumgart 胰肠吻合的前瞻性随机对照临床研究",探索本团队设计的改良 Blumgart 胰肠吻合技术能否在 LPD 的应用中真正做到简化手术步骤的同时保证较低的胰漏发生率。

## 参考文献:

- [1] 刘国华, 谭小宇, 戴东, 等. 改良Blumgart胰肠吻合在胰十二指肠切除术中的应用[J]. 中国普通外科杂志, 2020,29(3):276-283.
- [2] Cameron J L, Pitt H A, Yeo C J, et al. One hundred and forty-five consecutive pancreaticoduodenectomies without mortality[J]. Ann Surg, 1993,217(5):430-435, 435-438.
- [3] Gagner M, Pomp A. Laparoscopic pylorus-preserving pancreatoduodenectomy[J]. Surg Endosc, 1994,8(5):408-410.
- [4] Pedrazzoli S. Pancreatoduodenectomy (PD) and postoperative pancreatic fistula (POPF): A systematic review and analysis of the POPF-related mortality rate in 60,739 patients retrieved from the English literature published between 1990 and 2015[J]. Medicine (Baltimore), 2017,96(19):e6858.
- [5] Olakowski M, Grudzinska E, Mrowiec S. Pancreaticojejunostomy-a review of modern techniques[J]. Langenbecks Arch Surg, 2020,405(1):13-22.
- [6] Di Martino M, de la Hoz R A, Martin-Perez E. Blumgart pancreaticojejunostomy: does it

- reduce postoperative pancreatic fistula in comparison to other pancreatic anastomoses?[J]. Ann Transl Med, 2020,8(12):736.
- [7] Nagakawa Y, Takishita C, Hijikata Y, et al. Blumgart method using LAPRA-TY clips facilitates pancreaticojejunostomy in laparoscopic pancreaticoduodenectomy[J]. Medicine (Baltimore), 2020,99(10):e19474.
- [8] McMillan M T, Malleo G, Bassi C, et al. Defining the practice of pancreatoduodenectomy around the world[J]. HPB (Oxford), 2015,17(12):1145-1154.
- [9] 彭兵, 王昕, 蔡合. 胰肠吻合技巧及研究进展[J]. 中国普外基础与临床杂志, 2019,26(4):395-398.
- [10] Peng S Y, Wang J W, Lau W Y, et al. Conventional versus binding pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized trial[J]. Ann Surg, 2007,245(5):692-698.
- [11] Chen X P, Huang Z Y, Lau J W, et al. Chen's U-suture technique for end-to-end invaginated pancreaticojejunostomy following pancreaticoduodenectomy[J]. Ann Surg Oncol, 2014,21(13):4336-4341.
- [12] Grobmyer S R, Kooby D, Blumgart L H, et al. Novel pancreaticojejunostomy with a low rate of anastomotic failure-related complications[J]. J Am Coll Surg, 2010,210(1):54-59.
- [13] Oda T, Hashimoto S, Miyamoto R, et al. The Tight Adaptation at Pancreatic Anastomosis Without Parenchymal Laceration: An Institutional Experience in Introducing and Modifying the New Procedure[J]. World J Surg, 2015,39(8):2014-2022.
- [14] Hirono S, Kawai M, Okada KI, et al. Modified Blumgart Mattress Suture Versus Conventional Interrupted Suture in Pancreaticojejunostomy During Pancreaticoduodenectomy: Randomized Controlled Trial[J]. Ann Surg, 2019, 269(2):243–251. doi: 10.1097/SLA.00000000000002802.
- [15] Zhang XJ, Zhang W, Zhang T, et al. The safety and efficiency of the Blumgart anastomosis in pancreaticojejunostomy after pancreaticoduodenectomy[J]. Chinese Journal of Hepatobiliary Surgery, 2013, 19(11):831–835. doi:10.3760/cma.j.issn.1007–8118.2013.11.007.
- [16] Neychev VK, Saldinger PF. Minimizing shear and compressive stress during pancreaticojejunostomy: rationale of a new technical modification[J]. JAMA Surg, 2014, 149(2):203–207. doi: 10.1001/jamasurg.2013.2256
- [17] Sun P-J, Yu Y-H, Li J-W and Cui X-J .A Novel Anastomosis Technique for Laparoscopic Pancreaticoduodenectomy: Case Series of Our Center's Experience.Front. Surg. 8:583671. doi: 10.3389/fsurg.2021.583671.

[18] Poves I, Morató O, Burdío F, Grande L. Laparoscopic-adapted Blumgart pancreaticojejunostomy in laparoscopic pancreaticoduodenectomy. Surg Endosc. 2017 Jul;31(7):2837-2845. doi: 10.1007/s00464-016-5294-y. Epub 2016 Nov 1. PMID: 27804043.

### 2. 研究目的

传统 Blumgart 吻合的 LPD 手术为对照,评价本团队设计改良 Blumgart 胰肠吻合术在 腹腔镜胰十二指肠切除术中的应用效果,即探讨本团队设计改良 Blumgart 胰肠吻合所耗费 时间要比传统 Blumgart 胰肠吻合时间短;同时对于减少 LPD 术后患者 POPF 的发生率方面 该改良 Blumgart 胰肠吻合方式优于传统 Blumgart 胰肠吻合方式。

### 3. 研究对象

经影像学(上腹部 MRI、MRCP/CT/CTA)和或十二指肠超声内镜评估肿瘤可切除、无远处转移的初诊为壶腹周围癌的患者。

#### 3.1 入选标准

可根治性切除的 I-III 期低位壶腹周围癌患者为对象,并在入选时全部符合以下标准:

- 1) 年龄 18-80 岁;
- 2) 影像学(上腹部MRI、MRCP/CT/CTA)诊断为壶腹周围(十二指肠乳头、壶腹部、胆总管下段、胰头部)肿瘤性病变;
  - 3) 经MDT讨论评估肿瘤未侵犯大血管(SMA,CA,CHA/SMV,PV) 可切除;
  - 4) 十二指肠超声内镜下诊断为壶腹周围癌;
  - 5) 内镜下活检病理证实为癌(非必需);
  - 6) 术前分期为 T3N1 以内;
  - 7) 未发现远处转移证据者;
  - 8) 心肺及肝肾功能可耐受手术;
  - 9) 患者及家属能够理解并愿意参与本研究,提供书面知情同意。

#### 3.2 排除标准

入选时符合以下标准的患者需从本试验中排除:

- 1) 诊断合并其他部位恶性肿瘤;
- 2) ASA分级≥IV级和/或ECOG体力状态评分>2分;
- 3) 具有严重的肝肾功能、心肺功能、凝血功能障碍或合并严重的基础疾病不能耐受手

#### 术者:

- 4) 术前有感染未控制者;
- 5) 怀孕或哺乳期妇女;
- 6) 具有严重的精神疾病病史;
- 7) 有研究者认为的其他临床、实验室情况病人不宜参加该项试验。

#### 3.3 退出标准

以下退出研究的情况系由病人的非依从及非治疗本身原因所致。

- 1) 术中探查证实远处转移患者,包括肝脏、盆腔、腹膜等;
- 2) 术中探查证实肿瘤无法根治性切除,需要改行姑息性短路手术如:胆肠吻合的患者;
- 3) 术中因各种因素导致手术中转开腹或终止手术的患者。
- 4)入选研究后,患者因各种原因要求退出本研究队列者;
- 5)入选研究后因各种原因患者不能或不愿继续完成研究计划者。

如果患者退出试验,应在 CRF 表中记录患者退出的原因及时间。

## 4. 方案设计

本研究采用前瞻性、随机、开放、平行对照、优效性试验设计。

#### 5. 样本量估算及分组

#### 5.1 样本量估算

本研究为平行对照设计的临床研究,试验组为采取改良Blumgart吻合的LPD患者,对照组为采取传统Blumgart吻合的LPD患者,观察试验组患者术后POPF发生率是否低于对照组患者。根据既往文献报道以及本团队既往手术经验:估计试验组的术后POPF发生率约为6%,对照组的术后POPF发生率约为16%,试验组与对照组按1:1比例分组,按照优效性试验两组总样本率计算,优效界值 $\triangle$ =5%, $\alpha$ =0.05, $\beta$ =0.2(功效=80%),利用PASS11软件计算得到试验组和对照组所需要的最小样本量 $N_1$ = $N_2$ =67例,假定研究对象的失访率为10%,则需要样本量 $N_1$ = $N_2$ =67÷0.9≈75例,即总样本量为150例。

#### 5.2 患者编号和随机化分组

将患者数据输入电脑来获得一个受试者编号,所有受试者编号将为3位数,患者在研究过程中始终使用该编号,且不会被重新分配,患者编号分配后撤回知情同意或中止研究

的患者将会保留他们的初始编号。随机化使用分层区组随机化法进行分组,根据分层因素进行分层,然后再在层内进行区组随机化分组。由于本研究目的是要对比试验组与对照组的术后胰瘘的发生率,而目前比较公认的是术前影响胰瘘发生率的因素主要为胰腺质地及胰管直径,因此,将胰腺质地(硬,软)和胰管直径(≤3mm,>3mm)这两个重要的预后因素作为分层因素,使用区组随机(层内区组数目为 2,长度为 4)的方法进行分组。实现上述分层区组随机化的分组可以通过随机化工具或软件进行。

#### 6. 研究步骤或治疗方案

#### 6.1 术前筛选合格的受试者(患者)

- 1)患者入院后完善术前相关检查(血常规、肝肾功能、心肺功能、上腹部 CTA/MRI、MRCP/十二指肠超声内镜)
- 2) 符合入选标准且不符合排除标准的患者按随机化分组行改良 Blumgart 胰肠吻合的 LPD 手术组(试验组)或行传统 Blumgart 胰肠吻合的 LPD 手术组(对照组)。

#### 6.2 手术方案

- 6.2.1 试验组及对照组采用下述共同的 LPD 手术流程:
  - 1. 术前准备及麻醉方式 术前留置胃管、尿管及中心静脉通道;采用气管插管全麻的麻醉方式
  - 手术体位
     平卧位
  - 3. 手术步骤
- (1) 建立人工气腹及操作孔:于脐下做小切口,气腹针穿刺建立人工气腹并维持气压于 13~15mmHg,然后以 10 mm 穿刺器穿刺腹腔,经穿刺器放入 30°腹腔镜进行探查,排除腹膜及脏器表面转移。于腹腔镜明视下再作 4 个穿刺孔,分别位于两侧腋前线肋缘下 2 cm 及平脐腹直肌外缘; 5 个 Trocar 呈 V 形分布。右侧分别为 12 mm(平脐腹直肌外缘)及 5 mm Trocar 作为主、副操作孔,其中 12 mm Trocar 操作孔,可置入超声刀、切割闭合器、血管夹钳等器械;左侧两个均为 5 mm Trocar 作为助手操作孔。
- (2)解剖性探查:用超声刀切开胃结肠韧带,暴露胰腺;先沿胰腺下缘分离显露肠系膜上静脉,再沿胰腺上缘解剖显露肝总动脉、肝固有动脉、胃十二指肠动脉,清扫上述动脉旁淋巴结,肝总动脉旁淋巴结常规送冰冻切片检查;离断胃右动脉、胃十二指肠动脉,显露门静脉;沿肠系膜上静脉、门静脉前方贯通胰后隧道,置入系带悬吊。游离胆总管,

解剖胆囊三角,夹闭并离断胆囊动脉,将胆囊从胆囊窝中剥离,夹闭胆囊管,暂不离断,解剖游离胆总管,用血管吊带悬吊,暂不离断,以减轻胆汁污染。

- (3)标本切除及取出:根据从足端向头端、从前向后、从左向右的原则。在距 Treitz 韧带约 15 cm 处应用直线型切割闭合器(白订)切断空肠,用超声刀离断近端空肠系膜及十二指肠系膜。将游离后的近端空肠经肠系膜上血管后方推向右侧。应用直线型切割闭合器( 蓝订) 横断胃窦、胃体交界处,切除远端胃。在门静脉左侧胰腺预定离断处,用超声刀切断胰腺,胰腺断面确切止血。若见到胰管,采用剪刀离断胰管,易于胰肠吻合。采用 Kocher 切口,游离十二指肠及胰头部。提出经肠系膜上血管后方推向右侧的近端空肠,用超声刀沿肠系膜上动脉鞘右侧逐步完整离断胰腺钩突系膜(全系膜切除)。对肠系膜上动脉至胰腺钩突的分支及钩突至门静脉的属支,分别夹闭后离断。在胆囊管与胆总管汇合部上方切断肝总管,一般采用剪刀,并使前壁稍高于后壁,右侧稍低于左侧,以有利于腹腔镜下胆肠吻合。标本完全游离后,放入标本袋,将脐部穿刺孔扩大成绕脐半周切口,取出标本。将标本进行切缘标记,送冷冻切片检查,确保肝总管、胰颈、钩突切缘阴性。
- (4)消化道重建:采用 Child 式重建。首先将远端空肠经结肠后上提,行胰肠吻合。 之后在距胰肠吻合口 10 cm 处行胆肠吻合,最后再将残胃与胆肠吻合口下方约 45cm 处的空 肠作胃空肠吻合。
- ①胆肠吻合步骤:首先将空肠浆膜层与胆管周围组织缝合1针,使两者靠近;在空肠对系膜缘切开一个与胆管口直径相当的口,行胆管-空肠黏膜对黏膜吻合;再将肠管浆肌层与肝门板组织行间断缝合,以减少张力。
- ②胃肠吻合步骤:分别在预定吻合的空肠侧壁及残胃后壁开口,以直线型切割闭合器(蓝订)订合胃和空肠,共同开口以 3-0 可吸收线缝合关闭,缝合前须确定胃管处于胃肠吻合口附近。
- (5) 引流: 彻底冲洗腹腔,检查无活动性出血后,在胰肠吻合口和胆肠吻合口后方各置 1 根引流管,分别经原腋前线左右穿刺孔引出。
- 6.2.2 试验组的改良 Blumgart 胰肠吻合的方案
- (1) 胰腺断面予止血后 3-0 Prolene 线交叉贯穿 U 型缝合胰腺与空肠后缘浆肌层  $3\sim5$  针(图 1A);
- (2)于胰管内置入直径相仿的支架管,距空肠残端约 5 cm 的对系膜缘空肠用电凝钩戳一小口,外留约 3~5 cm 的支架管另一端置入从小口处置入空肠肠腔内,胰腺、空肠开口黏膜

与支架管之间潜在间隙予 4-0 Prolene 线各作一荷包缝合关闭并相互靠拢打结并固定支架管 (图 1B):

(3) 再次 3-0 Prolene 线交叉 U 型或 8 字缝合胰腺前壁与空肠前缘浆肌层  $3\sim5$  针(图 1C),完成改良 Blumgart 胰肠吻合。



图 1 改良 Blumgart 胰肠吻合示意图

## 6.2.3 对照组的传统 Blumgart 胰肠吻合的方案

- (1) 胰腺断面予止血后 3-0 Prolene 线间断贯穿 U 型缝合胰腺与空肠后缘浆肌层 3~5 针(图 2A),各 U 型缝合针暂不打结;
- (2)于胰管内置入直径相仿的支架管,距空肠残端约 5cm 的对系膜缘空肠用电凝钩戳一小口,外留约 3~5 cm 的支架管另一端置入从小口处置入空肠肠腔内,胰管与空肠开口予 4-0 Prolene 线间断缝合 4-6 针作胰管空肠黏膜缝合 (图 2B、图 2C);
- (3)将第一步留在胰腺前缘的 3-0 Prolene 针线作胰腺前壁与空肠浆肌层的缝合,完成传统 Blumgart 胰肠吻合(图 2D)。



图 2 传统 Blumgart 胰肠吻合示意图

#### 6.3 手术人员要求

胆胰亚专科中心团队固定的主刀及一助。主刀及一助均已具备丰富的开展LPD手术的 经验。

## 6.4 术后治疗方案

术后两组患者均常规予抗感染、保护胃黏膜、生长抑素、营养支持治疗。术后第3天拔除胃管以及尿管,嘱患者进食冷流质食物并且下床活动;术后第5天停用生长抑素,复查上腹部CTA观察腹腔内情况,其余治疗方案根据患者实际情况制定。术后第1、3、5、7天复查血常规、血生化、肝功能、血清淀粉酶与脂肪酶、引流液淀粉酶、C反应蛋白、降钙素原,记录内容包括复查的相关抽血指标、每天引流量以及引流液性质和淀粉酶含量、两组患者生化漏、B/C级胰瘘、胃瘫等并发症的发生情况、拔除引流管时间以及出院时间。

#### 6.5 手术后出院标准

患者一般情况良好,基本恢复正常饮食和肠道功能;体温正常,腹部检查无阳性体征;相关实验室检查结果基本正常;复查CTA腹腔内未见明显腹腔积液及其他异常情况;术后腹部切口愈合良好。

#### 7. 随访方案

- 1) 随访计划及内容:术后前3个月,每1个月返院随访一次。随访内容包括患者食欲、精神、大小便等情况;血常规、血淀粉酶、生化常规、肿瘤标记物(主要是CA199)、腹部CT/MRI、引流管引流量及腹水淀粉酶(带有腹腔引流管患者)等内容。胰瘘指标的评价在术后第1、3、5、7天至出院每隔3天评价1次,在出院后第1、2、3个月各评价1次;生活质量在术前、术后第1、2、3个月各评价1次。
  - 2)建立完整数据库,采用由专人负责的随访机制。
  - 3) 随访时间节点: 术后至出院前、术后1、2、3个月。
- 4)在院评估和返院随访的时间节点以外,由专门的术后随访医护人员采取电话、信件问卷、电子邮件等形式进行跟踪随访。

#### 8. 研究结果的评价指标

本研究旨在以腹腔镜下传统 Blumgart 胰肠吻合术作为对照,评价探讨本团队设计改良 Blumgart 胰肠吻合术在 LPD 中的应用价值即能否真正做到简化手术步骤的同时保证较低的 胰漏发生率。(即探讨本团队设计改良 Blumgart 胰肠吻合所耗费时间要比传统 Blumgart

胰肠吻合时间短;同时对于减少LPD术后患者POPF的发生率方面该改良Blumgart 胰肠吻合方式优于传统Blumgart 胰肠吻合方式。)

#### 8.1 主要评价指标: (疗效指标)

术后胰瘘(Postoperative pancreatic fistula, POPF)的发生率。

术后胰瘘(POPF)的定义为"胰腺导管系统和另一个上皮表面之间形成的富含胰腺来源酶液体的异常通道"。国际胰腺外科研究组(International Study Group on Pancreatic Surgery, ISGPS)2016 版关于 POPF 的诊断标准为"术后>3 d 时,引流液淀粉酶含量大于血清淀粉酶正常值上限的 3 倍,且与临床治疗预后相关"(详见附录)。

#### 8.2 次要评价指标: (疗效指标)

1) 围手术期情况:

详细记录术中胰肠吻合耗费时间(Pancreaticoje junostomy Time, PJ-time)、LPD 总手术时间、术中出血、术中中转率、术后 30 天内并发症等情况。具体记录内容包括:

- ①胰肠吻合耗费时间(PJ-time)
- ②LPD 总手术时间
- ③术中出血量
- ④术中中转率
- (5)腹腔感染发生率
- 6 术后出血发生率
- (7)胃排空延迟发生率

术后并发症按照Clavien-Dindo系统划分(详见附录)。下列情况被视为术后严重并发症:术后出血,需输血>4U红细胞;术后因并发症需急诊二次手术或介入治疗;严重感染;患者因手术原因死亡等,应在术后1个月内报告;

- 2) 术后恢复情况,具体记录内容包括:
- ①首次肛门排气时间
- ②恢复流质饮食时间
- (3)住院时间
- 4)拔除引流管时间

术后发生不良事件按照不良事件报告表进行登记,如为严重不良事件,请填写严重不良事件表,并请在24小时内临床试验组长、伦理委员会。并填写SAE报告表。

#### 3) 术后生活质量情况:

采用欧洲癌症研究与治疗组织所制定的生活质量(Quality of life QoL)调查量表: EORTC QoL C30量表(详见附录)。

#### 8.2 次要评价指标: (安全性指标)

术后 90 天内死亡发生率

### 9. 安全性评价:

### 9.1 获益

根据相关报道指出,壶腹周围癌在国内外的发病率均显现出上升趋势,在粤西地区范围内也有着相同的趋势,因此,需要行胰十二指肠切除术的患者也越来越多。目前,随着微创外科器械以及技术的进步,腹腔镜胰十二指肠切除术已广泛开展。但对于一些基层医院来说,腹腔镜下的吻合技术仍是需要克服的困难。本团队对传统 Blumgart 胰肠吻合方式进行改良,旨在保证低胰瘘率的前提下,简化胰肠吻合步骤并且缩短其所耗费时间,使整体手术时间得以缩短,有利于患者术后恢复。再者,不忘"立足于基层医院,回馈于基层医院"的初心,本团队希望相对简易而安全的腹腔镜下胰肠吻合技术能为更多基层医院普外科医师所掌握与应用,以便于更多基层医院能够顺利开展腹腔镜胰十二指肠切除术,给广大患者带来健康与希望。

#### 9.2 风险

- 1)无论是试验组还是对照组实施的 LPD 手术均有可能出现术后胰瘘、腹腔感染、腹腔 出血、胃排空延迟、胆瘘、肿瘤转移和复发等风险。受试者的相关检查与规定的定期复查 将同时进行并严格按照规范进行。
- 2) 回顾性分析了本团队既往已开展的传统和改良 Blumgart 胰肠吻合的 LPD 手术 20 例, 其术后胰瘘发生率较低,同时并无严重术后并发症的发生,术后 90 天内死亡率为零,已证 实该试验安全有效,风险可控。

#### 9.3 风险防范措施

#### 9.3.1 指导原则:

- ①预防为主:发现病例,及时报告,积极采取有效措施控制病情发展。
- ②依法管理:在临床试验的全过程中,贯彻执行相关法律法规,对出现的突发事件和不良事件,要及时报告,在整个控制和救治工作中实行依法管理,对于违法行为,依法追

#### 究法律责任。

- ③分级负责:在临床试验中,严格执行标准化操作规程,定期或不定期监查、督察整个过程,做到及时发现,及时救治。
- ④快速反应:建立预警和医疗救治快速反应,强化人力、物力、财力储备,增强应急处理能力,按照早期发现,及时报告,依靠科学,措施果断的原则,及时准确处置。 9.3.2 组织管理:
- ①领导机构:在院长领导下由医务处具体负责组织实施突发事件的处理工作。负责监督本院医务人员的医疗服务工作,检查医务人员的执业情况、接受投诉并向其提供咨询服务。配合并协调与之相关的争议和处理。
- ②指挥体系:将临床试验中受试者损害及突发事件纳入医院抢救和正常的医疗纠纷处理工作中。
- ③日常管理工作: 临床试验机构办公室为日常的业务管理部门, 具体负责临床试验的业务指导, 组织管理与质量控制, 监督检查, 并负责日常信息沟通与组织协调工作及突发事件的报告。
- ④参与人员: 各专业科室医、护、技专业技术人员、ICU救护专业人员以及心理卫生人员。

#### 9.3.3 防范措施:

- ①伦理委员会的保证:临床试验开始前,试验方案经伦理委员会审议同意并签署意见 后方能实施;临床试验进行期间,试验方案的任何修改均需经伦理委员会批准后方能执行; 试验中发生任何受试者损害及严重不良事件,需向伦理委员会报告。
- ②主要研究者的保证:临床研究项目负责人应具有本科以上学历和高级职称,有临床试验方案中所要求的专业知识和经验,熟悉申办者所提供的与临床试验有关的资料和文献,并有权支配进行该项试验所需要的人员和设备;具有处理不良事件的能力和及时上报事件的责任心。
- ③研究者的保证:熟悉不良事件报告程序的标准操作规程;临床试验开始前,各抢救设备和急救药品及时到位,确保出现受试者损害及突发事件时,受试者在第一时间得到救

治。

- ④对受试者的保证:受试者必须是自愿参加并且对研究项目有充分的了解;必须始终尊重受试者保护自身的权利;尽可能采取措施以尊重受试者的隐私、资料的保密,并将其身体和精神以及人格的影响减至最小;向受试者告知该项试验的各方面情况后,受试者自愿确认其同意参加临床试验的过程,须以签名和注明日期的知情同意书作为文件证明。
- ⑤机构的保证:建立健全质量保证体系:对主要研究者资格的保证;对各专业科室设施的保证;对临床试验方案的质量保证;对临床试验数据资料的质量控制;建立符合GCP管理规范的工作制度、设计规范、标准操作规程;制定受试者损害和突发事件应急预案:成立受试者损害和突发事件处理小组,保证医疗过程中出现受试者损害及突发事件后,受试者或患者得到及时处理;做好受试者损害与突发事件预防、现场控制、应急处理及其他物资和技术的准备与协调调度。

## 9.3.4 不良事件:

不良事件(AE)是指在临床诊疗活动中以及医院运行过程中,任何可能影响病人的诊疗结果、增加病人的痛苦和负担、并可能引发医疗纠纷或医疗事故,以及影响医疗工作的正常运行和医务人员人身安全的因素和事件。该事件不一定与这种治疗有因果关系。因此,不良事件可以是任何不良的和非预期的体征(包括异常的实验室发现)和症状,或者是与医学产品使用有时间上的相关性的疾病,无论是否认为与研究有关。

研究过程中出现的肿瘤进展或恶化(包括出现新的转移灶和因为疾病进展而引起的死亡)应作为疗效评价的一部分,不应报告为不良事件或严重不良事件。

在临床研究期间所发生的所有不良事件将在病例报告表(CRF)的不良事件页上报告。不良事件的严重程度将使用美国国家癌症研究所不良事件通用术语标准(4.0版) (CTCAEv4.0 (http://ctep.cancer.gov/reporting/ctc.html)进行分级并按照CRF 上的要求详细报告。若发生未包含在CTCAE v 4.0中的不良事件,将采用下列五级分制:

| 轻度 | 感觉不适但是并不影响正常的日常活动 |
|------|-------------------|
| 中度 | 不舒服程度足以减少或影响日常活动 |
| 重度 | 不能工作或不能进行正常的日常活动 |
| 危及生命 | 立即出现生命危险 |
| 死亡 | 与不良事件有关 |

#### 9.3.4.1 严重不良事件的定义

严重不良事件(SAE)是指在治疗过程中出现的符合下列某一标准的任何不良医学情况:

- (1)致命性(导致死亡;注意:死亡是后果,不是事件);
- ②危及生命(注意: "危及生命"是指在事件发生时患者立即有死亡的危险,并不是指如果事件更严重一些的话会引起死亡这样的假设);
  - ③导致患者住院治疗或者住院时间延长;
  - (4)导致终身的或严重的残疾/功能缺陷;
  - (5)导致先天畸形或出生缺陷;
  - (6)在医学上具有重要意义或需要干预措施以防止上述任何一种后果的发生;

#### 9.3.4.2 因果关系

应使用下列标准评估不良事件与治疗的关系:

- 1)很可能有关:该类别指以很高程度的确定性认为与临床研究相关的不良事件。如果具备以下标准,可认为一个不良事件"很可能有关":
  - 不良事件的出现与手术具有合理的时间相关性。
- ②已知的患者疾病状态、环境或毒性因素或患者使用的其他治疗不能合理解释不良事件。
- 2)可能有关(必须有前两项):该类别指与本次研究不太可能有关,但是又不能肯定排除关联性的不良事件。如果具备以下标准,可认为一个不良事件"可能相关":
  - (1)不良事件的出现与手术具有合理的时间相关性。
- ②不良反应可能是由患者的疾病状态、环境或毒性因素或患者使用的其他合并治疗造成的。
  - 3) 可能无关(必须具有前两项): 该类别适用于满足下述标准的不良事件:
  - 不良事件的出现与手术不具有合理的时间相关性。
- ②不良事件明显由患者的疾病状态、环境或毒性因素或患者使用的其他合并治疗造成。
- 4) 无关:该类别指清楚明确地判断为仅由外部因素(疾病、环境等)引起,而且不符合"可能无关"、"可能有关"或"很可能有关"项下手术相关性判断标准的不良事件。

必须遵照ICH对临床试验安全性数据管理指南、快速报告的定义和标准进行。

#### 9.3.4.3 预期不良事件

手术相关不良事件:

本研究中试验组与对照组均需要建立气腹,特有的并发症包括:皮下气肿、高碳酸血症、穿刺并发的血管和胃肠道损伤、气体栓塞等。

LPD 手术共有并发症,主要有:

- 1) 胰瘘
- 2) 腹腔内活动性出血;
- 3) 消化道出血;
- 4) 吻合口出血; (包括胆道吻合口、胰肠吻合口、胃肠吻合口)
- 5) 吻合口瘘、淋巴漏;
- 6) 肠粘连、肠梗阻;
- 7) 内疝;
- 8) 结肠、脾脏等周围脏器损伤;
- 9) 切口并发症(感染、积液、裂开、愈合不良等);
- 10) 肺炎、泌尿系感染、肾功能衰竭、肝功能衰竭、心脑血管事件(包括血栓、栓塞等);
  - 11) 其他。

#### 9.3.4.4 不良事件处理措施

- 1) 根据具体情况采取必要的治疗措施,决定是否中止临床试验。并将其症状体征或实验室检查结果、出现时间、持续时间、程度、处理措施、经过等详细记录于病案,评价其与临床试验的相关性,由研究者签名并注明日期。
- 2) 发现不良事件时,研究者应立即处理并向科室负责人、伦理委员会及临床研究中心,根据病情决定必要的诊断与治疗措施,决定是否中止临床试验。所有不良事件件都应追踪调查,详细记录处理经过及结果,直到妥善解决或病情稳定,若化验异常者应追踪至恢复正常。追踪随访方式可根据不良反应的轻重选择住院、门诊、家访、电话、通讯等方式。
- 3) 不良事件的报告:在研究期间,不论患者接受哪种治疗,所发生的任何严重不良事件或是严重的实验室检查结果异常,研究者必须填写不良事件报告表和CFDA严重不良事件报告表,并在获悉后24 小时内报告给项目负责人、伦理委员会及临床研究中心。

SAE 报告联系人:广东医科大学附属医院肝胆胰二区办公室

单位联系人: 翟景威(广东医科大学附属医院)

手机: 18814103880

邮箱: 466269963@qq.com

地址:广东省湛江市霞山区人民大道南57号

- 4)记录:研究者应在原始病案和CRF表中记录受试者的症状、体征、实验室检查,损害出现的时间、持续时间、程度、处理措施和经过等,保证记录真实、准确、完整、及时、合法,填写严重不良事件报告表,签名并注明日期;在原始记录中应记录时间、报告方式以及报告的机构。
- 5) 随访: 研究者应对所有受试者损害进行随访,根据病情决定随访时间,在随访过程中给予必要的处理和治疗措施,以确保将受试者损害降至最低,充分保证受试者安全。详细记录随访的经过和处理的结果。
- 9.3.5 突发事件处理措施:

A、突发公共卫生事件处理措施:

- (a)报告:在正常工作日,当班医护人员应立即报告受试者损害突发事件处理小组,节假日或夜间应立即报告行政总值班,由总值班向受试者损害和突发事件处理小组报告,小组人员应综合评估,初步判断突发公共卫生事件的性质,并向上级行政部门报告,提出是否启动突发公共卫生事件应急预案的建议。
- (b) 启动应急预案: 经上级卫生行政部门批准后,启动突发公共卫生事件应急预案,包括: ★成立特殊门诊、急诊及留诊室。
- ★院领导值班:院办迅速制定院领导值**班表**,保证一名院领导24小时值班,全面负责突发事件;医务处每日有专门人员24小时值班;所有相关人员24小时手机开通,确保联络畅通,并于每日上午8:00、下午5:00到院部汇总相关信息,集中讨论,处理有关问题。
- ★保障物质供应:紧急调集人员、储备相关物资、交通工具以及相关的设施、设备,确保 医疗资源的合理配置,保障重点科室的医疗应急物资供应。
- ★疏散或隔离:根据病情需要,必要时对人员进行疏散和隔离。
- ★救援与记录: 医务人员严格遵守防护措施,对患者进行紧急医疗救护和现场救治;书写详细、完整的病历记录;需要转送他院的,按照规定转送至接诊的或指定的医疗机构。
- ★培训和演练: 平时针对突发公共卫生事件的性质进行应急处理相关知识、技能的培训和

演练, 随时做好应急准备工作。

B、自然灾害的处理措施:

火灾、水灾和地震等发生应立即与"119"或"110"联系,并通知受试者损害和突发事件处理小组,节假日或夜间应立即报告总值班,由总值班通知上述小组。小组负责人立即向院长报告,接受指示,同时由院办向全院通告紧急状况。相关职能部门做好各自工作。

C、紧急停电、停水处理措施:

处理措施:一旦由于局部线路的原因造成科室突然停电,医护人员应当立即电话通知总务 科管理人员,后勤管理人员在接到通知后立即安排专业人员赶赴现场紧急抢修线路,尽快恢复供电。各科室提前接到停水、停电通知,务必提前安排好工作;避开该时间段进行的相关检查或治疗。对于临床试验方案中要求必须当天检测的标本,应确保标本质量的前提下妥善保存,待供水或供电恢复后再行检测。

- 9.3.6 处罚: 医务人员有下列行为之一的,由医院有关部门责令改正、通报批评、给予警告;对科室负责人和其他直接责任人依法给予降级或撤职的纪律处分;造成受试者(患者)致残、死亡或疾病传播、流行或者对社会公众健康造成其他严重危害后果,构成犯罪的,依法追究刑事责任。
  - (1)未按规定履行不良事件或突发事件报告职责,隐瞒、缓报或者谎报的;
  - ②未按规定对受试者出现的不良事件或突发事件及时采取措施的;
  - ③突发事件来临时拒绝接诊病人的;
  - (4)突发事件来临时拒不服从医院工作调度的。
- 10. 招募过程(包括招募程序及启动时间、招募材料、预期招募人数)
- **10.1 招募程序:**包括招募受试者、筛选合格受试者、获得受试者的知情同意三个环节。 10.1.1 招募受试者
- 受试者招募工作人员:负责接诊的医生、分管的住院医师、也可以是临床监管医生。 招募人员确定后开始制定招募计划与需求。
- 招募方式:第一种是招募人员确定该患者符合试验要求,推荐患者参加试验;第二种 是患者的主治医生不是试验的研究者,确定患者符合临床试验要求,询问患者意愿后与研 究者联系纳入患者。

- 招募的场所: 医院门诊, 住院部或者健康体检中心。
- 接待潜在受试者:设置专门的招募窗口由专人负责接待来访的受试者或者利用专线电话对咨询患者进行疑问解答。
- 按纳入和排除标准以及医生的临床经验初步判断受试者入选可能性。
- 受试者合格性筛查:对初步判断可能合格的受试者进行试验概况说明,进行体格检查或实验室检查,根据检查结果,再次确认受试者是否真正符合试验纳入排除标准。
- 受试者知情同意:对筛查合格的患者进行临床试验方案的详细说明,并告知可能存在的获益和风险,做到充分知情。

#### 10.1.2 筛选合格受试者

将对初步判断可能合格的受试者进行合格性判断,事先应当根据合格性标准,设计好单独的、清晰明确的病历筛查表。合格性判断标准就是把临床试验的诊断标准、纳入排除标准进行细化为可判断的条目,并根据疾病和试验设计情况排除特殊人群(如妊娠、传染性疾病)和患有相关并发症的患者。通过合格性判断标准判断受试者是否符合临床试验的要求,符合研究条件的患者进入临床试验,判断不合格的受试者予以剔除,不对其进行入组。不符合要求的患者产生的额外判断费用应由研究项目承担,并给予常规治疗。具体的合格性判断流程如下:①根据事先确定的诊断标准纳入符合标准的受试者;②再根据事先确定的纳入标准纳入符合标准的受试者;③最后根据排除标准将具有排除标准特征的患者排除纳入不具有排除标准特征的患者。

#### 10.1.3 获得受试者的知情

通过合格性筛查后,研究人员应该对每一个受试者进行知情同意告知并确认签字。

#### 10.2 启动时间

项目获得审批通过并通过伦理委员会批准后开始启动受试者招募。

#### 10.3 招募材料

知情同意书。

#### 10.4 预期招募人数

符合入选条件的200名拟行腹腔镜胰十二指肠切除术的壶腹周围癌患者。

#### 10.5 研究对象参加研究的时间(每次参与时间与总时间)

入组并已接受本试验规定手术到出院为研究对象第一次参加研究时间;手术后3个月返院到完善相关检查;总的参加研究时间为手术后3个月结束。

## 11、数据管理与统计分析计划

#### 11.1 数据处理

## 11.1.1 数据收集

所有资料均应及时、如实、详细地纪录在病历登记表(Case Report Form, CRF)或CRF软件中。研究者必须按照方案要求将信息输入CRF,研究中心委派监督员将检查CRF的完整性和准确性,并指导研究中心人员进行必需的修改或补充。CRF由地区监督员送交数据处理,一份复件保留在研究中心,一份附件则作为监督员的工作附件。CRF将交与可靠的医学数据处理员进行数据录入。病历记录表应由各本单位指派专人填写并经各单位该项目负责人签名后方能视为有效病例。

临床试验结束后,按临床总结规范要求写出临床分总结报告。

#### 11.1.2 病例报告表 (CRF)

在临床试验中,需要将规定的观察或检查项目记录在病例报告表中。

病例报告表中的内容须与原始资料完全一致,对于由原始资料计算所得的结果,其计算的 依据应可以溯源。

在填写时须符合以下标准:

- (1) 用黑色签字笔或黑色圆珠笔填写;
- (2)已经签署知情同意书并符合入选标准的病例,即使没有进行药物治疗或治疗后判定为 不符合入选标准,也应填写病例报告表。
- (3)进行修正时,须用横线划去原记录(不能用修正液等修改),但要保证原记录的可辨认, 并在更正处签名并签署更正日期。
- (4) 对于未查项目, 须标注 "ND(Not Done)"。

#### 11.1.3 数据库管理与质量控制

CRF内的数据项目将使用具有二次录入审核的复式输入法输入研究数据库。文本项目 (如注释)从CRF输入一次之后只能手动核对。随后,数据管理人员使用从确认程序和数 据库列表中打印的错误信息,对输入数据库的信息进行系统检查。如有必要,一个独立的 文件对DQF(Data Quality Form)处理及归档进行试验特殊操作有明确说明(如确认计划)。数据库在宣告完成并且无误后将被锁定。在那以后任何对数据库的改动只能经由获得临床研究领导者、研究统计学家和数据管理者联合书面同意而实现。结果的判读由不知道患者分组情况的第三方进行,确保结果的客观性。

#### 11.2 统计分析

## 11.2.1 分析人群定义:

入组并进行手术治疗的病人构成本次试验的意向性治疗人群(ITT intention-to-treat, population)和遵从本临床试验方案要求并完成本次研究的病人构成符合临床实验的方案人群(PP-Per Protocol),统计分析将采用CFLO(Carry Forward Of the Last Observation)方法对缺失数据处理。

#### 11.2.2 统计分析方法

- 1)根据分析指标的性质确定统计学描述和统计学检验的分析方法。对连续型变量分析分布范围、均数、中位数、标准差和四分位数间距,两组比较连续性变量采用τ检验或非参数检验;对分类变量列表分析其发生例数和发生率,两组分类变量采用χ2检验、Fisher's精确概率法或列连表资料统计分析方法。不论在任何阶段,均采用概率P值进行统计推断,统计学显著性差异界值用0.5。关于安全性数据统计分析计划,所有的安全性参数都以列表和总结表的形式进行描述。不良事件和实验室参数根据NCI CTCAE v4.0标准进行评估。研究分析的安全性数据包括:报告的所有不良事件和严重不良事件(无论其相关性如何)的发生率。
- 2)非劣效检验的相关统计分析方法。在针对有效性的统计分析过程中,采用可信区间法,因此,对于本非劣效检验主要效应指标为低优指标时,若试验组措施与对照组措施胰瘘发生率差异的双侧95%可信区间的上限小于事先设定的判断界值△时,则可判定非劣效性假设成立,若上述非劣效结论成立,即可进行优效性检验,若试验组措施与对照组措施胰瘘发生率差异的双侧95%可信区间的上限小于事先设定的判断界值-△时,则优效结论成立,研究结论可判定为非劣效且优效。

#### 12、资料保密计划

参加试验及在试验中的个人资料均属保密。可以识别受试者身份的信息将不会透露给研究小组以外的成员,除非获得受试者的许可。所有的研究成员和研究申办方都被要求对受试者的身份保密。受试者的档案将保存在有锁的档案柜中,仅供研究人员查阅。为确保
研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅受试者的个人资料。这项研究结果发表时,将不会披露受试者个人的任何资料。

### 13、伦理要求与知情同意

### 13.1 取得伦理委员会批件

在研究机构启动临床试验之前,必须获得研究机构伦理委员会的批件。在试验进行中研究者应按要求提交试验进度报告给伦理委员会,试验结束后还应该书面报告伦理委员会。

## 13.2 知情同意

在病例登记前,主要研究者或研究者按照知情同意书向受试者说明临床试验相关内容等,随后给予受试者足够的时间考虑,并由受试者自主决定是否签署知情同意书。主要研究者或研究者以及受试者在知情同意书上签名并注明日期(说明日期、获得知情同意日期)。若试验相关人员进行补充说明,则该试验相关人员也须签名或填写姓名并盖章并记录说明日期。另外,试验过程中若因试验方案发生变更,或获得有可能影响受试者继续参加试验的新信息而需修订知情同意书时,则需向受试者说明变更的内容,并由受试者再次自主决定是否签署新的知情同意书。如果受试者不同意签署新的知情同意书,则受试者须中止临床试验。知情同意书一式两份,原件由中心保存、复印件由受试者保留。

## 13.3 知情同意书的修订

主要研究者可以依据最新的信息考虑修改知情同意书,新修订的知情同意书必须经过 伦理委员会的审批同意后,才能在临床试验中使用。已经签署了旧的知情同意书且没有完 成临床试验的患者,在继续进行试验之前应再次签署新的知情同意书,新、旧版本的知情 同意书均须保留做原始资料。

#### 13.4 受试者的隐私保护

在病例报告表、统计分析报告、临床试验报告、不良事件报告中,凡涉及到患者信息的内容均不得出现患者的真实信息。患者可通过编号和姓名缩写进行辨别。

## 13.5 研究方案的修改

本方案经伦理委员会批准后,若在实施过程中有重大修改,由临床研究负责人撰写"方案修改说明书",并签字,同时需报请伦理委员会批准后方可实施。未做原则性修改,由临床研究小组、统计学家、方法学家共同讨论决定并签字。

## 14、质量控制和质量保证

### 14.1 数据管理

所有入选病例必须由主管医生完成CRF表的填写,CRF表中所有项目均须完成。所填写的项目不得涂改,如需修改,应先将填错的数据用一短横线划掉,然后在其上方填上正确的结果,并在旁边签名和注明修改日期。主管医生在填写完成后应认真检查核对所有CRF中数据,并在CRF表中签名,表明已检查过,务必保证数据填写的真实性、准确性。完成的CRF表由监察员审查后进行保管,进行数据录入与管理工作。

#### 14.2 本研究的治疗控制

控制内容:指标的填写是否有遗漏,是否与原始资料一致,是否准确填写。常见问题:不同医生填写一致性不高;填写缺失、错误、与研究病例不一致。

解决方法:在本研究开始前,参与研究的医生与人员必须经过统一的培训,统一记录方式与判断标准。确认评价指标的一致性、可靠、完整及准确。在研究过程中,由PI指派的监察员定期对研究进行监查访问及审核,以保证研究方案中的所有内容得到严格遵守、填写CRF的正确以及填写数据的真实性、准确性。

### 14.3 原始资料的保存

本研究的原始资料包括已签署的知情同意书、有关实验室及影像学检查报告、病例记录及其他相关记录等均应保存于广东医学院附属医院档案室。

#### 14.4 试验盲法的设置

本研究因为手术方式不同,无法进行设盲,但对随访人员和疗效评估人员进行设盲,即疗效评估人员在不知道患者具体分组的情况下进行疗效评估及随访数据资料的收集,以消除主观因素对研究结果的影响,尽量减少研究偏倚。

#### 15. 数据和记录的保存

研究者有责任确保研究记录不会受到意外损坏;受试者的医疗记录应贴上明确的标签,以确保防止因错误意外销毁文件。研究者及研究机构须保存临床试验相关资料到临床试验结束后五年,作为医疗文件的原始资料按照医院的有关规定保存,但不得少于临床试验结束后五年。

## 16. 研究流程

所有受试者必须是经影像学(上腹部 MRI、MRCP/CT/CTA)和或十二指肠超声内镜评估肿瘤可切除、无远处转移的初诊为壶腹周围癌的患者,并且进行临床分期。合纳入标准,不属于排除标准者均为潜在受试者。经过 MDT 讨论可行 LPD 手术的患者,术前由主治医师对受试者和家属进行告知,解释两种术式的差异,征求受试者本人和家属的意见,是否同意随机分组。同意随机分组的患者签署知情同意书后,纳入本研究进行随机分组并接受术后随访。(见附录 1)

## 17. 总结报告和论文发表

- 1) 临床研究完成研究总结后可发表论文、参加国内外学术会议。
- 2) 本研究成果以论文形式公开发表。预计发表SCI论文1-2篇。

## 试验流程



## 评估时间表及流程

| 阶段 | | | 随访阶段 | | |
|---|---|---|---|---|---|
| 项目 | 术前 | 术后-出<br>院前 | 术后1月 | 术后2月 | 术后3月 |
| 病史病历,基本资料 | $\sqrt{}$ | | | | |
| 术前抽血项目 | √ | | | | |
| 术前常规检查项目 | $\sqrt{}$ | | | | |
| 生活质量量表术前基线值 | $\checkmark$ | | | | |
| 围手术期安全性 | | $\sqrt{}$ | | | |
| 手术记录(术中出血、手术总时间、<br>胰肠吻合时间等) | | V | | | |
| 病理评估 | | $\sqrt{}$ | | | |
| 术后抽血: 术后第1、3、5、7天;<br>7天后3天复查一次。 | | V | √ | V | V |
| 术后引流管引流液生化、淀粉酶 | | $\sqrt{}$ | 引流管未<br>拔除者(√) | 引流管未<br>拔除者(√) | |
| 术后恢复情况:恢复排气时间、恢<br>复流质饮食时间 | | V | | | |
| 术后随访 | | | V | V | √ |
| 肿瘤标记物(CA199等) | V | √ | V | V | <b>V</b> |
| 上腹部 CT 增强或 CTA | $\sqrt{}$ | V | V | | |
| 生活质量问卷 | V | | V | V | V |
| 分析漏缺项目、失访患者 | √ | $\sqrt{}$ | V | V | V |

## 备注:

术前抽血项目包括:血常规等血液分析、生化全套、肿瘤标记物如 CA199 等;

术前常规检查包括:心肺功能评估;上腹部 CTA 或 MRI 增强;

十二指肠超声内镜等。

术后抽血检查项目: 血常规、血清淀粉酶、降钙素原、生化、

肝肾功能、肿瘤标记物如 CA199 等。

## ASA 分级标准

指美国麻醉师协会(ASA)于麻醉前根据病人体质状况和对手术危险性进行分类, 将病人分成的六级。

第一级: 体格健康,发育营养良好,各器官功能正常。围手术期死亡率 0.06%-0.08%;

第二级:除外科疾病外,有轻度并存病,功能代偿健全。围手术期死亡率 0.27%-0.40%;

第三级:并存病情严重,体力活动受限,但尚能应付日常活动。围手术期死亡率1.82%-4.30%;

第四级:并存病严重,丧失日常活动能力,经常面临生命威胁。围手术期死亡率 7.80%-23.0%;

第五级:无论手术与否,生命难以维持24小时的濒死病人。围手术期死亡率9.40%-50.7%;

第六级:确证为脑死亡,其器官拟用于器官移植手术。

第一、二级病人麻醉和手术耐受力良好,麻醉经过平稳。第三级病人麻醉有一定危险,麻醉前准备要充分,对麻醉期间可能发生的并发症要采取有效措施,积极预防。第四级病人麻醉危险性极大,即使术前准备充分,围手术期死亡率仍很高。第五级为濒死病人,麻醉和手术都异常危险,不宜行择期手术。

# ECOG 体力状态评分标准

| 级别 | 功能状态 | 相当于Karnofsky评分 |
|----|-------------------------------------------|----------------|
| 0 | 活动能力完全正常,与起病前活动能力无任何差异。 | 90- 100 |
| 1 | 能自由走动及从事轻体力活动,包括一般家务或办公室工作,但 不能从事较重的体力活动。 | 70-80 |
| 2 | 能耐受肿瘤的症状,能自由走动及生活自理,己丧失工作能力,但白天卧床时间不超过50% | 50-60 |
| 3 | 肿瘤的症状严重,白天卧床或坐轮椅时间超过50%,但还能起床站立,仅部分生活自理 | 30-40 |
| 4 | 病重卧床不起, 生活不能自理。 | 10-20 |
| 5 | 死亡 | 0 |

# 附录5 随机化申请表

申请日期: 年 月 日 随机号:

| 一般资料 | | |
|---------------------|-------------|--------------------------|
| 姓名缩写: | 年龄:岁 | 性别: 男□ 女□ |
| 体重: Kg | 身高: m | BMI指数: Kg/m <sup>2</sup> |
| 临床分期: cT□ N□ M0( 期) | | |
| 病理类型: ●肠型腺癌 ●胰胆管型 | 以腺癌 ●其他类型(行 | 行穿刺有病理的填写) |

| 入选标准核对表 | | |
|--------------------------------------------------|---|---|
| 入选标准 | 是 | 否 |
| 1.性别不限;年龄介于18-75岁 | | |
| 2. 影像学(上腹部MRI、MRCP/CT/CTA)和十二指肠超声内镜诊断为壶腹周围肿瘤性病变; | | |
| 3. 经MDT讨论评估肿瘤未侵犯大血管(SMA,CA,CHA/SMV,PV)可切除; | | |
| 4.术前十二指肠超声内镜病理活检证实为壶腹周围癌; | | |
| 5.未发现远处转移证据者; | | |
| 6.术前分期为T3N1以内; | | |
| 7.具备足够的器官功能; | | |
| 8.病人或家属,能够理解研究方案并愿意参与本研究,提供书面知情同意。 | | |
| 以上各条标准必须全部为"是",否则患者无法入组。 | | |

应用改良 Blumgart 胰肠吻合技术的腹腔镜胰十二指肠切除术治疗壶腹周围癌的前瞻性、开放、随机、平行对照临床研究

| 排除标准核对表 | | |
|----------------------------------|---|---|
| 排除标准 | 是 | 否 |
| 1. 近期诊断合并其他部位恶性肿瘤; | | |
| 2. ASA分级≥IV级和/或ECOG体力状态评分>2分; | | |
| 3.具有严重的肝肾功能、心肺功能、凝血功能障碍或合并严重的基础疾 | | |
| 病不能耐受手术者; | | |
| 4.具有严重的精神疾病病史; | | |
| 5.怀孕或哺乳期妇女;; | | |
| 6.术前有感染未控制者; | | |
| 7.有研究者认为的其他临床、实验室情况病人不宜参加该项试验。 | | |
| 以上各条标准必须全部为"否",否则患者无法入组。 | | |

是否符合入组: 是□ 否□ 未入组原因

符合入组者随机化结果: A 组□ B 组

# 附录 6 AJCC 壶腹癌分期标准(2018 年 第八版)

#### 原发肿瘤(T)

- Tx 原发肿瘤无法评价
- To 无原发肿瘤证据
- Tis 原位癌
- T<sub>1a</sub> 肿瘤局限于 Vater 壶腹或 Oddi 括约肌
- Тıь 肿瘤超出 Oddi 括约肌和/或侵及十二指肠黏膜下
- T2 肿瘤侵及十二指肠固有肌层
- T3a 肿瘤侵及胰腺 (≤0.5cm)
- T3b 肿瘤侵及胰腺>0.5cm,或者胰腺周围软组织/十二指肠浆膜,无腹腔动脉和肠系膜上动脉侵袭
- T4 肿瘤侵及腹腔动脉, 肠系膜上动脉, 和/或肝总动脉, 无论肿瘤大小

#### 区域淋巴结(N)

- N<sub>x</sub> 区域淋巴结无法评估
- N<sub>0</sub> 无区域淋巴结转移
- N<sub>1</sub> 有 1-3 个区域淋巴结转移
- N<sub>2</sub> 有 4 个以上区域淋巴结转移

#### 远处转移(M)

- M<sub>0</sub> 无远处转移
- M<sub>1</sub> 有远处转移

解剖分期/预后组别

| Stage | T | N | M |
|-------|----------|--------------|-------|
| 0 | Tis | $N_0$ | $M_0$ |
| I | $T_1$ | $N_0$ | $M_0$ |
| I A | $T_{1b}$ | $N_0$ | $M_0$ |
| IΒ | $T_2$ | $N_0$ | $M_0$ |
| II A | $T_{3a}$ | $N_0$ | $M_0$ |
| IIB | $T_{3b}$ | $N_0$ | $M_0$ |
| IIIA | $T_{1a}$ | $N_0$ | $M_0$ |
| | $T_{1b}$ | $N_1/N_{1c}$ | $M_0$ |
| | $T_2$ | $N_{2a}$ | $M_0$ |
| | $T_{3a}$ | $N_1/N_{1c}$ | $M_0$ |
| | $T_{3b}$ | $N_{2a}$ | $M_0$ |
| IIIB | $T_4$ | Any N | $M_0$ |

应用改良 Blumgart 胰肠吻合技术的腹腔镜胰十二指肠切除术治疗壶腹周围癌的前瞻性、开放、随机、平行对照临床研究

| | Any T | $N_2$ | $M_0$ |
|----|-------|-------|-------|
| IV | Any T | Any N | $M_1$ |

## 注: 1.cTNM 是临床分期, pTNM 是病理分期

2.Tis 包括肿瘤细胞局限于腺体基底膜(上皮内)或黏膜固有层(黏膜内),未穿过黏膜肌层到达黏膜下层。

## ISGPS 术后胰瘘(POPF)的定义及分级系统(2016版)

2016版术后胰瘘分级临床评定表

| | | | 100 1 11110 112 | | | |
|---|---|---|---|---|---|---|
| | 引流液淀粉酶含量力<br>血清淀粉酶正常值上限 | | 胰周持续<br>引流>3周 | 临床相关的胰瘘<br>治疗措施改变 <sup>2)</sup> | 经皮或内镜下<br>穿刺引流 | 血管造影介人治疗术后<br>胰瘘相关出血 |
| BL(非术后胰瘘) | 是 | | 否 | 否 | 否 | 否 |
| B级术后胰瘘" | 是 | | 是 | 是 | 是 | 是 |
| C级术后胰瘘" | 是 | | 是 | 是 | 是 | 是 |
| | 二次手术 | 术后胰瘘 | 相关的感染征象 | 术后胰瘘相 | 关器官衰竭" | 术后胰瘘相关死亡 |
| BL(非术后胰瘘) | 否 | 否 | | 7 | 5 | 否 |
| B级术后胰瘘 <sup>1)</sup> | 否 | 是,但未 | 出现器官衰竭 | 7 | § | 否 |
| C级术后胰瘘" | 是 | 是,出现 | <b>见器官功能衰竭</b> | 夷 | Ē | 是 |

注:1)临床相关的术后胰瘘被定义为引流液淀粉酶含量大于血清淀粉酶正常值上限的3倍且发生了与术后胰瘘直接相关的临床状态及预后改变2)表示住院或重症监护室停留时间延长,包括采取治疗胰瘘的一些相关措施。包括使用生长抑素类似物、完全肠内或肠外营养、输注血制品或其他药物治疗3)术后器官衰竭被定义为呼吸功能障碍发展到需要再插管,肾功能不全发展到需要血液透析,心功能不全发展到需要使用强心药物



注:1)术后胰瘘相关事件

图 1 2016 版术后胰瘘的临床发生发展流程图

## 术后并发症 Clavien-Dindo 系统分级

I: 术后出现不需要药物、外科、内镜以及放射介入等治疗并发症,但包括: 止吐药、退烧药、止痛药、利尿药、电解质、理疗; 床边敞开的切口感染也归于此类

Ⅱ: 需要 I 期并发症以外药物治疗: 包括输血和全肠外营养;

Ⅲ: 需要外科、内镜、放射介入等干预

Ⅲa: 干预不需要全身麻醉

Ⅲb: 干预需要全身麻醉

IV: 威胁生命的并发症(包括中枢神经系统并发症)需要入住 ICU

**Ⅳa:** 一个器官功能不全(包括透析)

IVb: 多器官功能不全

V: 死亡

## 国际生命质量(EORTC QLQ C30)问卷

#### 亲爱的患者:

疾病的发生会给人带来一系列生理及心理的变化,包括身体上的各种客观和主观的不适,个人的自尊和自信心受挫,个人社会功能难以得以实现,生存质量受到严重影响。在生物-心理-社会医学这一现代医学模式指引下,我们不仅关注疾病本身,更关注您的生活和生命的质量。当前国际上有各种生命质量评估的量表,不同的量表所适用的疾病、评估的效力有所不同。我们现选择这份 EORTC QLQ C30 量表评估您个人的实际情况,请您认真填写,我们将会把您回馈的结果用于指导您疾病的治疗。

请您指出过去一段时间内对以下症状或问题的程度,选择最符合您的项目。问题的答案没有对错,您只需告诉我们您最真实的感受。

| 完全没有 | 有一点 | 相当多 | 非常多 |
|---|---|---|---|
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| 完全没有 | 有一点 | 相当多 | 非常多 |
| 1 | 2 | 3 | 4 |
| 完全没有 | 有一点 | 相当多 | 非常多 |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| 1 | 2 | 3 | 4 |
| | 1 1 1 1 1 1 2 2 2 3 1 1 1 1 1 1 1 1 1 1 | 1 2 | 1 2 3 |

应用改良 Blumgart 胰肠吻合技术的腹腔镜胰十二指肠切除术治疗壶腹周围癌的前瞻性、开放、随机、平行对照临床研究

| 20. | 您集中精力做事有困难吗,如读报纸或看电视? | 1 | 2 | 3 | 4 |
|-----|-----------------------|---|---|---|---|
| 21. | 您觉得紧张吗? | 1 | 2 | 3 | 4 |
| 22. | 您觉得忧虑吗? | 1 | 2 | 3 | 4 |
| 23. | 您觉得脾气急躁吗? | 1 | 2 | 3 | 4 |
| 24. | 您觉得压抑(情绪低落)吗? | 1 | 2 | 3 | 4 |
| 25. | 您感到记忆困难吗? | 1 | 2 | 3 | 4 |
| 26. | 您的身体状况或治疗影响您的家庭生活吗? | 1 | 2 | 3 | 4 |
| 27. | 您的身体状况或治疗影响您的社交活动吗? | 1 | 2 | 3 | 4 |
| 28. | 您的身体状况或治疗使您陷入经济困难吗? | 1 | 2 | 3 | 4 |

对下列问题,请在1-7之间选出一个最适合您的数字并画圈。

您如何评价在过去一星期内您总的健康情况? 1234567 (从左往右为非常差到非常好) 您如何评价在过去一星期内您总的生活质量? 1234567 (从左往右为非常差到非常好)

感谢您的参与!